CLINICAL TRIAL: NCT00129922
Title: Phase III Study to Compare 6 Courses of FEC (Fluorouracil, Epirubicin and Cyclophosphamide) vs. 4 Courses of FEC Followed by 8 Weekly Paclitaxel Administrations, as Adjuvant Treatment for Node Positive Operable BC Patients
Brief Title: Fluorouracil, Epirubicin, and Cyclophosphamide Alone or Followed by Paclitaxel for Early Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Spanish Breast Cancer Research Group (Other)
Collaborators: Bristol-Myers Squibb (Industry); Pfizer (Industry); Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEICAM 9906
Record Dates: First submitted 2005-08-10; First posted 2005-08-12 (Estimated); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer
Keywords: Axillary node positive breast cancer.; Sequential drug administration.; Weekly paclitaxel.
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; Fluorouracil; Epirubicin; Cyclophosphamide

ARMS (2):
- Fluorouracil+Epirubicin+Cyclophosphamide (Active Comparator): 5-FU+4-Epirubicin+Cyclophosphamide
  Interventions: Drug: Fluorouracil; Drug: Epirubicin; Drug: Cyclophosphamide
- FEC followed by Paclitaxel (Experimental): 5-FU+4-Epirubicin+Cyclophosphamide
  Interventions: Drug: paclitaxel; Drug: Fluorouracil; Drug: Epirubicin; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: paclitaxel
  Other Names: Taxol
  Arms: FEC followed by Paclitaxel
Drug: Fluorouracil
  Other Names: 5-FU
Drug: Epirubicin
  Other Names: 4-Epirubicin
Drug: Cyclophosphamide

SUMMARY:
The efficacy of adjuvant chemotherapy is limited in patients with a high risk of recurrence.

Also, for axillary positive node patients, optimum chemotherapy regimens are still under discussion. Some previous studies suggest that, in the subset of node-positive patients, treatments based on sequential administration of anthracyclines and taxanes are more efficient. Paclitaxel dose-dense (weekly) administration renders an improved therapeutic index (activity/toxicity).

The study is designed to compare 6 courses of FEC scheme (600/90/600), a combination of proven efficacy in node positive breast cancer patients, versus 4 FEC courses followed by 8 weekly paclitaxel administrations (100mg/m2).

The study hypothesis is that 5-year disease-free survival in the control arm will be 60%. The investigators expect to increase this by 8% with the experimental treatment. With an alpha error of 0.05, 80% power, and a post-randomization estimated drop-out rate of 10%, 1250 patients are needed, 625 per arm.

DETAILED DESCRIPTION:
The primary endpoint of study-5-year disease-free survival (DFS) will be assessed by Kaplan Meier analysis. Secondary endpoints included overall survival and analysis of the prognostic and predictive value of clinical and molecular markers. Associations and interactions will be assessed with a multivariable Cox proportional hazards model for DFS for the following covariates: age, menopausal status, tumor size, lymph node status, type of chemotherapy, tumor size, positive lymph nodes, HER2 status, and hormone receptor status. All statistical tests will be two-sided.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Histological diagnosis of breast cancer.
* Node positive operable breast cancer (stages II-III).
* Breast cancer surgery, consisting of radical mastectomy or conservative surgery, plus lymphadenectomy with at least 6 extirpated nodes. Surgery must have happened in the 8 weeks prior to randomisation.
* Age >=18 and <= 70 years old.
* Negative pregnancy test. Adequate contraceptive method during the study participation.
* Performance status of 90-100 (Karnofsky index) or ECOG <=1.
* Haemoglobin >= 10 g/dl; neutrophils > 1,500/cc; platelets > 100,000/cc.
* Adequate hepatic function with bilirubin, SGOT and SGPT < 1.5 x upper normal limit (UNL).
* Adequate cardiac function documented by left ventricular ejection fraction (LVEF).
* Adequate renal function with creatinine < 1.5 mg/dl.

Exclusion Criteria:

* Previous chemotherapy, hormone therapy and/or radiotherapy for breast cancer.
* Bilateral breast cancer. Lobular in situ carcinoma.
* Previous or current malignancies, except for basal skin carcinoma, cervical in situ carcinoma or superficial bladder carcinoma, adequately treated.
* History of arrhythmias and/or congestive heart failure or cardiac blocking grade 2-3; history of myocardial infarction in 6 months before recruitment.
* Inability for treatment and study compliance.
* Pregnant or lactating women.
* Active infection.
* History of hypersensitivity to cremophor or cyclosporine.
* Pre-existing grade 2 motor or sensorial neurotoxicity (National Cancer Institute Common Toxicity Criteria [NCI CTC]).
* Hormonal receptor status not determined.
* Any other criteria which, in investigator's opinion, may jeopardize patient's security or compliance.
* Administration of other investigational product in the 30 days prior to randomisation; current participation in another clinical trial.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1289 (Actual)
Dates: Start 1999-11 (Actual); Primary Completion 2005-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
disease-free survival | 5 years
  From the date of randomization of each patient included to the 1st documented evidence of recurrence

SECONDARY OUTCOMES:
Overall survival | From date of randomization until the date of death from any cause, assessed up to 100 months
  Overall survival will be measured from the day of randomization to the date of death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Hospital General Universitario de Elche; Study Director, Study Director — Hospital Universitario Marqués de Valdecilla; Study Director, Study Director — Hospital Provincial de Córdoba
Locations (64):
- Spain (64):
  - Hospital Universitario Virgen de los Lirios, Alcoy, Alicante
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital General Universitario de Elda, Elda, Alicante
  - Hospital Municipal de Badalona, Badalona, Barcelona
  - Hospital Unviersitario Germans Trias i Pujol, Badalona, Barcelona
  - Althaia-Xarxa Assistencial de Manresa, Manresa, Barcelona
  - Corporació Sanitaria Parc Taulí, Sabadell, Barcelona
  - Hospital Espíritu Santo, Santa Coloma de Gramenet, Barcelona
  - Hospital Universitario Mutua de Terrassa, Terrassa, Barcelona
  - Consorci Sanitari de Terrassa, Terrassa, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital de Jerez de la Frontera, Jerez de la Frontera, Cádiz
  - Hospital Universitario Puerto Real, Puerto Real, Cádiz
  - Onkologikoa, Donostia / San Sebastian, Gupúzcoa
  - Hospital Donostia, Donostia / San Sebastian, Gupúzcoa
  - Hospital de Barbastro, Barbastro, Huesca
  - Hospital Universitario de Gran Canaria Dr. Negrín, Las Palmas de Gran Canaria, Las Palmas
  - Complejo Hospitalario Universitario Insular-Materno Infantil, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital Universitario de Móstoles, Móstoles, Madrid
  - Hospital Clínico Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital de Cabueñes, Gijón, Principality of Asturias
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Hospital Universitario San Joan de Reus, Reus, Tarragona
  - Hospital de la Ribera, Alzira, Valencia
  - Hospital de Sagunto, Sagunto, Valencia
  - Hospital Universitario Cruces, Barakaldo, Vizcaya
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Centro Oncológico de Galicia, A Coruña
  - Hospital General Universitario de Alicante, Alicante
  - Hospital del Mar, Barcelona
  - Clínica Oncológica Corachán, Barcelona
  - Hospital Clinic i Provincial, Barcelona
  - Hospital Universitario Puerta del Mar, Cadiz
  - Hospital General Universitario de Ciudad Real, Ciudad Real
  - Hospital Provincial de Córdoba, Córdoba
  - Hospital General Universitario de Guadalajara, Guadalajara
  - Hospital Juan Ramón Jiménez, Huelva
  - Complejo Hospitalario de Jaén, Jaén
  - Hospital de León, León
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Clínico Universitario San Carlos, Madrid
  - Hospital Clínico Unviersitario Virgen de la Victoria, Málaga
  - Hospital General Universitario Morales Meseguer, Murcia
  - Complejo Hospitalario de Ourense, Ourense
  - Hospital Rio Carrión, Palencia
  - Hospital Unviersitario de Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Virgen de la Salud, Toledo
  - Hospital Provincial de Toledo, Toledo
  - Hospital Universitario La Fe, Valencia
  - Instituto Valenciano de Oncología, Valencia
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Universitario Arnau de Vilanova de Valencia, Valencia
  - Hospital Universitario Dr. Peset, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid
  - Hospital Provincial de Zamora, Zamora
  - Hospital Clínico Universitario de Zaragoza "Lozano Blesa", Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza
  - Hospital de Txagorritxu, Vitoria-Gasteiz, Álava

REFERENCES:
- [Result] Martin M, Rodriguez-Lescure A, Ruiz A, Alba E, Calvo L, Ruiz-Borrego M, Santaballa A, Rodriguez CA, Crespo C, Abad M, Dominguez S, Florian J, Llorca C, Mendez M, Godes M, Cubedo R, Murias A, Batista N, Garcia MJ, Caballero R, de Alava E. Molecular predictors of efficacy of adjuvant weekly paclitaxel in early breast cancer. Breast Cancer Res Treat. 2010 Aug;123(1):149-57. doi: 10.1007/s10549-009-0663-z. PMID 20037779
- [Result] Ebbert MT, Bastien RR, Boucher KM, Martin M, Carrasco E, Caballero R, Stijleman IJ, Bernard PS, Facelli JC. Characterization of uncertainty in the classification of multivariate assays: application to PAM50 centroid-based genomic predictors for breast cancer treatment plans. J Clin Bioinforma. 2011 Dec 23;1:37. doi: 10.1186/2043-9113-1-37. PMID 22196354
- [Result] de la Haba-Rodriguez J, Rodriguez-Lescure A, Ruiz A, Alba E, Calvo L, Carrasco E, Escudero MJ, Martin M. Regional and seasonal influence in patient's toxicity to adjuvant chemotherapy for early breast cancer. Breast Cancer Res Treat. 2011 Jan;125(1):273-8. doi: 10.1007/s10549-010-1136-0. Epub 2010 Aug 28. PMID 20803065
- [Result] Bastien RR, Rodriguez-Lescure A, Ebbert MT, Prat A, Munarriz B, Rowe L, Miller P, Ruiz-Borrego M, Anderson D, Lyons B, Alvarez I, Dowell T, Wall D, Segui MA, Barley L, Boucher KM, Alba E, Pappas L, Davis CA, Aranda I, Fauron C, Stijleman IJ, Palacios J, Anton A, Carrasco E, Caballero R, Ellis MJ, Nielsen TO, Perou CM, Astill M, Bernard PS, Martin M. PAM50 breast cancer subtyping by RT-qPCR and concordance with standard clinical molecular markers. BMC Med Genomics. 2012 Oct 4;5:44. doi: 10.1186/1755-8794-5-44. PMID 23035882
- [Result] Pajares B, Pollan M, Martin M, Mackey JR, Lluch A, Gavila J, Vogel C, Ruiz-Borrego M, Calvo L, Pienkowski T, Rodriguez-Lescure A, Segui MA, Tredan O, Anton A, Ramos M, Camara Mdel C, Rodriguez-Martin C, Carrasco E, Alba E. Obesity and survival in operable breast cancer patients treated with adjuvant anthracyclines and taxanes according to pathological subtypes: a pooled analysis. Breast Cancer Res. 2013 Nov 6;15(6):R105. doi: 10.1186/bcr3572. PMID 24192331
- [Result] Martin M, Prat A, Rodriguez-Lescure A, Caballero R, Ebbert MT, Munarriz B, Ruiz-Borrego M, Bastien RR, Crespo C, Davis C, Rodriguez CA, Lopez-Vega JM, Furio V, Garcia AM, Casas M, Ellis MJ, Berry DA, Pitcher BN, Harris L, Ruiz A, Winer E, Hudis C, Stijleman IJ, Tuck DP, Carrasco E, Perou CM, Bernard PS. PAM50 proliferation score as a predictor of weekly paclitaxel benefit in breast cancer. Breast Cancer Res Treat. 2013 Apr;138(2):457-66. doi: 10.1007/s10549-013-2416-2. Epub 2013 Feb 20. PMID 23423445
- [Result] Prat A, Cheang MC, Martin M, Parker JS, Carrasco E, Caballero R, Tyldesley S, Gelmon K, Bernard PS, Nielsen TO, Perou CM. Prognostic significance of progesterone receptor-positive tumor cells within immunohistochemically defined luminal A breast cancer. J Clin Oncol. 2013 Jan 10;31(2):203-9. doi: 10.1200/JCO.2012.43.4134. Epub 2012 Dec 10. PMID 23233704
- [Result] Martin M, Brase JC, Calvo L, Krappmann K, Ruiz-Borrego M, Fisch K, Ruiz A, Weber KE, Munarriz B, Petry C, Rodriguez CA, Kronenwett R, Crespo C, Alba E, Carrasco E, Casas M, Caballero R, Rodriguez-Lescure A. Clinical validation of the EndoPredict test in node-positive, chemotherapy-treated ER+/HER2- breast cancer patients: results from the GEICAM 9906 trial. Breast Cancer Res. 2014 Apr 12;16(2):R38. doi: 10.1186/bcr3642. PMID 24725534
- [Result] Cheang MC, Martin M, Nielsen TO, Prat A, Voduc D, Rodriguez-Lescure A, Ruiz A, Chia S, Shepherd L, Ruiz-Borrego M, Calvo L, Alba E, Carrasco E, Caballero R, Tu D, Pritchard KI, Levine MN, Bramwell VH, Parker J, Bernard PS, Ellis MJ, Perou CM, Di Leo A, Carey LA. Defining breast cancer intrinsic subtypes by quantitative receptor expression. Oncologist. 2015 May;20(5):474-82. doi: 10.1634/theoncologist.2014-0372. Epub 2015 Apr 23. PMID 25908555
- [Result] Martin M, Brase JC, Ruiz A, Prat A, Kronenwett R, Calvo L, Petry C, Bernard PS, Ruiz-Borrego M, Weber KE, Rodriguez CA, Alvarez IM, Segui MA, Perou CM, Casas M, Carrasco E, Caballero R, Rodriguez-Lescure A. Prognostic ability of EndoPredict compared to research-based versions of the PAM50 risk of recurrence (ROR) scores in node-positive, estrogen receptor-positive, and HER2-negative breast cancer. A GEICAM/9906 sub-study. Breast Cancer Res Treat. 2016 Feb;156(1):81-9. doi: 10.1007/s10549-016-3725-z. Epub 2016 Feb 24. PMID 26909792
- [Result] Templeton AJ, Rodriguez-Lescure A, Ruiz A, Alba E, Calvo L, Ruiz-Borrego M, Santaballa A, Rodriguez CA, Crespo C, Ramos M, Gracia-Marco JM, Lluch A, Alvarez I, Casas MI, Sanchez-Arago M, Caballero R, Carrasco E, Amir E, Martin M, Ocana A; GEICAM 9906 Study Investigators. Prognostic role for the derived neutrophil-to-lymphocyte ratio in early breast cancer: a GEICAM/9906 substudy. Clin Transl Oncol. 2018 Dec;20(12):1548-1556. doi: 10.1007/s12094-018-1885-5. Epub 2018 May 15. PMID 29766456
- [Result] Sestak I, Martin M, Dubsky P, Kronenwett R, Rojo F, Cuzick J, Filipits M, Ruiz A, Gradishar W, Soliman H, Schwartzberg L, Buus R, Hlauschek D, Rodriguez-Lescure A, Gnant M. Prediction of chemotherapy benefit by EndoPredict in patients with breast cancer who received adjuvant endocrine therapy plus chemotherapy or endocrine therapy alone. Breast Cancer Res Treat. 2019 Jul;176(2):377-386. doi: 10.1007/s10549-019-05226-8. Epub 2019 Apr 30. PMID 31041683
- [Result] Camp NJ, Madsen MJ, Herranz J, Rodriguez-Lescure A, Ruiz A, Martin M, Bernard PS. Re-interpretation of PAM50 gene expression as quantitative tumor dimensions shows utility for clinical trials: application to prognosis and response to paclitaxel in breast cancer. Breast Cancer Res Treat. 2019 May;175(1):129-139. doi: 10.1007/s10549-018-05097-5. Epub 2019 Jan 23. PMID 30673970
- [Result] Ethier JL, Ocana A, Rodriguez Lescure A, Ruiz A, Alba E, Calvo L, Ruiz-Borrego M, Santaballa A, Rodriguez CA, Crespo C, Ramos M, Gracia Marco J, Lluch A, Alvarez I, Casas M, Sanchez-Arago M, Carrasco E, Caballero R, Amir E, Martin M. Outcomes of single versus double hormone receptor-positive breast cancer. A GEICAM/9906 sub-study. Eur J Cancer. 2018 May;94:199-205. doi: 10.1016/j.ejca.2018.02.018. Epub 2018 Mar 21. PMID 29573665
- [Derived] Martin M, Carrasco E, Rodriguez-Lescure A, Andres R, Servitja S, Anton A, Ruiz-Borrego M, Bermejo B, Guerrero A, Ramos M, Santaballa A, Munoz M, Cruz J, Lopez-Tarruella S, Chacon JI, Alvarez I, Martinez P, Miralles JJ, Polonio O, Jara C, Aguiar-Bujanda D. Long-term outcomes of high-risk HR-positive and HER2-negative early breast cancer patients from GEICAM adjuvant studies and El Alamo IV registry. Breast Cancer Res Treat. 2023 Sep;201(2):151-159. doi: 10.1007/s10549-023-07002-1. Epub 2023 Jun 20. PMID 37338729
- See also: Click here for more information about this study: GEICAM 9906 — http://www.geicam.org